CLINICAL TRIAL: NCT05510596
Title: Contribution of Magnetic Resonance Imaging in Immune Effector Cell-Associated Neurotoxicity Syndrome
Brief Title: Magnetic Resonance Imaging in Immune Effector Cell-Associated Neurotoxicity Syndrome
Acronym: MR-ICANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL20_0424
Record Dates: First submitted 2022-06-03; First posted 2022-08-22 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, B-Cell; Neurotoxicity
Keywords: Neurotoxicity; CAR-T CELLS; Immune cells associated neurotoxicity syndrome; Cytokine release syndrome
MeSH Terms: conditions — Lymphoma, B-Cell; Neurotoxicity Syndromes; Cytokine Release Syndrome | interventions — Magnetic Resonance Spectroscopy; Contrast Media; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with CAR-T Cell treatment (Other): Single arm All patient will undergo an MRI with contrast injection, a blood withdrawal and a neurological consultation with neuropsychological tests
  Interventions: Other: Magnetic Resonance Imaging with contrast injection; Other: Blood withdrawal; Other: Neuropsychological tests

INTERVENTIONS:
Other: Magnetic Resonance Imaging with contrast injection — Magnetic Resonance Imaging with contrast injection
Other: Blood withdrawal — Blood withdrawal : serum, plasma, cytokine assay
Other: Neuropsychological tests — Neuropsychological tests

SUMMARY:
The treatment of large-cell B-cell lymphomas refractory to more than 2 lines of therapy has recently been revolutionized by the use of immunotherapies consisting of autologous genetically modified cells or CAR-T CELLS (chimeric antigen receptor-T cells), which very significantly increase progression-free survival and overall survival. Nevertheless, this therapy is frequently associated with cytokine release syndrome and in approximately 20% to 60% of patients with neurological complications that can sometimes be dramatic and are associated with a significant mortality rate.

The mechanisms behind this neurotoxicity are unclear.

Despite the frequent occurrence of neurological toxicity characterized in particular by headache, tremor, and encephalopathy that is most often transient, brain imaging by CT or, preferably, MRI are most often normal. The rare abnormalities that have been identified suggest the presence of cytotoxic edema associated with the existence of transient modifications of the blood-brain barrier.

To date, the management of neurotoxicity associated with CAR-T CELLS remains empirical. It combines early management of cytokine release syndrome (by administration of anti-IL6) and treatment with corticosteroids, the objective of which would be to control neurotoxicity more specifically. A better understanding of the pathophysiological mechanisms associated with this neurotoxicity appears essential today in order to be able to propose adapted prevention and treatment methods.

Main objectives are to compare tissue permeability by quantitative MRI measurement of Ktrans to the theoretical peak of neurotoxicity between patients with CAR-T Cell-induced neurotoxicity and those without neurotoxicity and to Study, by MRI, the evolution of tissue microcirculatory parameters (from D-3 to D7) between groups of patients with or without the occurrence of neurotoxicity associated with CAR-T CELL treatment.

For this purpose, 25 subjects will be included (the investigators hypothesize 40% with treatment-induced neurological impairment).

DETAILED DESCRIPTION:
The treatment of large-cell B-cell lymphomas refractory to more than 2 lines of therapy has recently been revolutionized by the use of immunotherapies consisting of autologous genetically modified cells or CAR-T CELLS (chimeric antigen receptor-T cells), which very significantly increase progression-free survival and overall survival. Nevertheless, this therapy is frequently associated with cytokine release syndrome and in approximately 20% to 60% of patients with neurological complications that can sometimes be dramatic and are associated with a significant mortality rate.

The mechanisms behind this neurotoxicity are unclear but may include :

* A "systemic" toxicity associated with the cytokine release syndrome. This toxicity would thus be favoured by the associated inflammatory response syndrome manifested in particular by hyperthermia, changes in blood pressure, and an increase in CRP, ferritin and the number of white blood cells.
* A breakdown of the blood-brain barrier, as evidenced by increased protein levels, cellularity and cytokine levels in the cerebrospinal fluid. Among other things, this rupture could be promoted by the synthesis of proinflammatory cytokines (IL6, TNF-alpha, IFN-gamma) that would promote endothelial activation.
* Direct toxicity to neurons and/or microglial cells.

Despite the frequent occurrence of neurological toxicity characterized in particular by headache, tremor, and encephalopathy that is most often transient, brain imaging by CT or, preferably, MRI are most often normal. The rare abnormalities that have been identified suggest the presence of cytotoxic edema associated with the existence of transient modifications of the blood-brain barrier.

To date, the management of neurotoxicity associated with CAR-T CELLS remains empirical. It combines early management of cytokine release syndrome (by administration of anti-IL6) and treatment with corticosteroids, the objective of which would be to control neurotoxicity more specifically. A better understanding of the pathophysiological mechanisms associated with this neurotoxicity appears essential today in order to be able to propose adapted prevention and treatment methods.

Objectives:

Main:

* To Compare tissue permeability by quantitative MRI measurement of Ktrans to the theoretical peak of neurotoxicity between patients with CAR-T Cell-induced neurotoxicity and those without neurotoxicity.

Secondary:

* To Study, by MRI, the evolution of tissue microcirculatory parameters (from D-3 to D7) between groups of patients with or without the occurrence of neurotoxicity associated with CAR-T CELL treatment.
* To Correlate the values of the MRI parameters with the usual clinical and biological parameters known to be associated with the occurrence of neurotoxicity (at D0 and theoretical peak).
* To Correlate the values of the MRI parameters with the values (at D0 and at NADIR) of a panel of cytokines of interest (V-PLEX Neuroinflammation Panel Human 1 Kit, Meso Scale Discovery®).

ELIGIBILITY:
Inclusion Criteria:

* Subject aged from 18 years old
* Subject able to understand the nature, purpose and methodology of the study
* Subject with diffuse large B-cell lymphoma to be treated with axicabtagene ciloleucel, tisagenlecleucel or brexucabtagene autoleucel for their lymphoma.

Exclusion Criteria:

* Refusal to sign the informed consent
* Subject presenting a cerebral localization of his lymphoma
* Contraindication to the realization of an MRI (metallic foreign body, pace-maker, cochlear implants)
* Claustrophobic subject
* Subject with a neurodegenerative disease (Parkinson's, Alzheimer's...)
* Subject with psychiatric disorders such as psychosis, except for anxiety-depressive episodes
* Subject with a systemic pathology with neurological manifestation
* Subject with a previous or evolving neurological pathology
* Subject with or with a history of severe head trauma (group 2 or 3 according to the Masters classification)
* Contraindication to the use of gadoline contrast products (severe renal insufficiency, liver transplantation, known or suspected hypersensitivity to the product)
* Pregnant or breastfeeding women
* Patient under tutelage
* Patient under curatorship
* Patient deprived of liberty
* Not a beneficiary of a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Study of tissue permeability evolution | 10 days
  Quantitative measurement of KTRANS (rate of contrast agent transfer from plasma to the extravascular extracellular space, reflecting capillary permeability).
  (Time in second)

SECONDARY OUTCOMES:
Qualitative analysis of tissue signals | 10 days
  FLAIR hypersignals analysis by MRI (signal of a tissue superior to the signal of the surrounding tissues) (visual assessment)
Qualitative analysis | 10 days
  Microbleeding analysis (3DEPI T2*)
Qualitative analysis | 10 days
  Analysis of contrast on injected 3DT1 MRI
Semi-quantitative analysis of parameters associated with permeability | 10 days
  Wash-in, Wash-out (Time in second)
Semi-quantitative analysis of parameters associated with permeability | 10 days
  Time to peak (TPP) (Time in second)
Semi-quantitative analysis of parameters associated with permeability | 10 days
  AUC (area under the curve shows blood volume) (SI x Time)
Quantitative analysis of parameters associated with permeability | 10 days
  Kep: rate of return transfer of the contrast agent from the extravascular extracellular space to the plasma (Volume/Time/Volume)
Quantitative analysis of parameters associated with permeability | 10 days
  Ve: volume fraction of the extravascular space (Percentage %)
Quantitative analysis of parameters associated with permeability | 10 days
  Vp: volume fraction of the plasma space. (Percentage %)
Quantitative analysis | 10 days
  Cerebral blood flow analysis (3DPCASL) (L/min)
Quantitative analysis | 10 days
  Cerebral volumetric analysis (3DT1) (cm3)
Quantitative analysis | 10 days
  Diffusion coefficient (ADC) (mm²/s)
Quantitative analysis | 10 days
  Perfusion factors (perfusion fraction f) (Percentage %)
Quantitative analysis | 10 days
  Perfusion factors (pseudo-diffusion D* at the microvascular compartment) (x10^-3 mm²/s)
Qualitative analysis : comparison with clinical data | 10 days
  Presence, absence of neurotoxicity and inflammation
Comparison with biological data from standard care and "Neuroinflammation Panel Human 1 Kit" | 10 days
  Comparison of MRI data with biological markers (such as CRP, ferritin, white blood cell count, LDH, procalcitonin, fibrinogen) and cytokine profile of neuroinflammation by multiplex immunoassay kit. An ultrasensitive multiplex using electrochemiluminescence.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse CARRA-DALLIERE, Dr, Principal Investigator — Montpellier University Hospital
Locations (1):
- Neurology department, Montpellier University Hospital, Montpellier, Occitanie, France